CLINICAL TRIAL: NCT07386678
Title: Study of Imaging and Molecular Biomarkers in Uncomplicated Rhegmatogenous Retinal Detachment
Acronym: Cohort-NHS
Status: Not yet recruiting | Type: Observational
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: EDGE 179423
Record Dates: First submitted 2026-01-27; First posted 2026-02-04 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Retinal Detachment Rhegmatogenous; Proliferative Vitreoretinopathy; Proliferative Vitreoretinopathy in Rhegmatogenous Retinal Detachment
Keywords: Cytokines; Imaging
MeSH Terms: conditions — Vitreoretinopathy, Proliferative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples Without DNA — Vitreous
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Disease or general study area: Uncomplicated rhegmatogenous retinal detachment (RRD) and risk of proliferative vittroretinopathy (PVR)

Purpose and nature of the study:

1. Characterise the cytokine profile of vitreous fluid in uncomplicated RRD.
2. Develop a risk model to predict development of PVR after retinal detachment surgery using imaging and molecular biomarkers.
3. To develop deep learning/artificial intelligence (AI) models for PVR detection in retinal detachment.

Inclusion criteria:

50 adult ( ≥18 years) patients with uncomplicated rhegmatogenous retinal detachments without PVR.

What participating will involve:

Pre- and post-operative assessments and intervention will follow standard of care for patients with rhegmatogenous retinal detachments.

Additional intervention will include non-invasive imaging of anterior chamber flare, vitreous, wide-field retina, macula optical coherence tomography (OCT) and macula OCT-angiography (OCT-A) as well as, seeking participant's consent on collecting their vitreous fluid at time of their surgery for cytokine analysis.

DETAILED DESCRIPTION:
This is an observational cohort study of 50 participants with uncomplicated rhegmatogenous retinal detachment. Participants will have their vitreous fluid collected at the time of surgery for cross-sectional analysis of cytokine milieu and a series of pre-operative and post-operative non-invasive imaging over 3 months. Unfortunately, 15-20% of the patients with primary retinal detachment will have recurrent retinal detachments following surgery secondary to an anomalous scarring process called proliferative vitreoretinopathy (PVR).

Therefore, aims of this study are to:

1. Characterise the cytokine profile of vitreous fluid in uncomplicated RRD.
2. Develop a risk model to predict development of PVR after retinal detachment surgery using imaging and molecular biomarkers.
3. To develop deep learning/artificial intelligence (AI) models for PVR detection in retinal detachment.

Above will guide future treatments for PVR and further identify high risk populations not just from a clinical perspective but with the utilisation of their imaging and molecular biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years
* Uncomplicated primary rhegmatogenous retinal detachment
* PVD present
* No PVR-A/B/C
* Phakic or pseudophakic.

Exclusion Criteria:

* Patients <18 years
* Patients lacking capacity
* Previous vitrectomy
* Previous cryopexy
* Aphakia
* No fundal view
* Diabetic retinopathy of any severity
* Retinal detachment secondary to infective causes e.g. acute retinal necrosis, toxoplasmosis scars
* Retinal detachment secondary to congenital defects e.g. optic disc pit/coloboma
* Exudative retinal detachment
* Tractional retinal detachment
* Ongoing involvement in another ocular trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Adults ≥18 years
  * Uncomplicated primary rhegmatogenous retinal detachment
  * Moorfields Eye Hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-03-02 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Characterise the cytokine milieu in an uncomplicated RRD eye. | 3 months
  Study cytokine profile using a multiplex assay that includes all relevant cytokines.

SECONDARY OUTCOMES:
Develop a risk model for development of PVR after retinal detachment surgery using imaging and molecular biomarkers. | 3 months
  Study demographics, existing and novel risk factors from imaging aqueous, vitreous, retinal vasculature and retinal structure, and cytokine molecular biology. Use a risk model for risk-stratification of patients who develop PVR re detachment.
To develop deep learning AI models for PVR detection in retinal detachment. | 3 months
  Using ultra-widefield retinal imaging and optical coherence tomography in human retinal detachment models.

CONTACTS AND LOCATIONS:
Locations (1):
- Moorfields Eye Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Cytokine profile
Supporting Information: Study Protocol, ICF